CLINICAL TRIAL: NCT02110615
Title: MA Childhood Obesity Research Demonstration (CORD) Project
Brief Title: Mass in Motion Kids in the Clinical Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Massachusetts Department of Health (Other Government); Harvard School of Public Health (HSPH) (Other); National Initiative for Children's Healthcare Quality (Unknown); Texas Institute for Measurement, Evaluation and Statistics (Unknown); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elsie Taveras, MD, Chief, Division of General Academic Pediatrics, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5U18DP003370 (NIH)
Record Dates: First submitted 2014-04-02; First posted 2014-04-10 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Primary Care Practice Changes (Experimental): The clinical intervention components included (1) advanced training on clinical quality improvement and obesity prevention, assessment, management; (2) computerized, point-of-care decision support tools for clinicians; (3) implementation of multi-disciplinary weight management programs within the community health centers, e.g. Healthy Weight Clinics (HWC); (4) integrating community health workers into the primary care and HWC teams; and (5) health center environmental changes to support behavior change modification.
  Interventions: Other: Primary Care Practice Changes

INTERVENTIONS:
Other: Primary Care Practice Changes — The clinical intervention components included (1) advanced training on clinical quality improvement and obesity prevention, assessment, management; (2) computerized, point-of-care decision support tools for clinicians; (3) implementation of multi-disciplinary weight management programs within the community health centers, e.g. Healthy Weight Clinics (HWC); (4) integrating community health workers into the primary care and HWC teams; and (5) health center environmental changes to support behavior change modification.

SUMMARY:
Mass in Motion Kids is a whole-of-community intervention in Fitchburg and New Bedford, Massachusetts that incorporates evidence-based interventions across multiple sectors and at multiple levels. The overall goal of the study is to examine the extent to which the comprehensive, systematic intervention reduces childhood obesity among underserved children.

The clinical intervention implements evidence-based interventions each city's federally-qualified community health center. Intervention components aim to improve primary and secondary prevention of childhood obesity and implement changes at four levels: clinician; parent-family; organizational; and environmental. We additionally provide training and educational materials to other pediatric clinicians in the two communities. The clinical intervention components include (1) advanced training on clinical quality improvement and obesity prevention, assessment, management; (2) computerized, point-of-care decision support tools for clinicians; (3) implementation of multi-disciplinary weight management programs within the community health centers, e.g. Healthy Weight Clinics (HWC); (4) integrating community health workers into the primary care and HWC teams; and (5) health center environmental changes to support behavior change modification.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-12 years
* Patient of the community's federally qualified health center

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3765 (Actual)
Dates: Start 2011-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline Body Mass Index at 2 years | 2 years prior to intervention start through study end (expected average of 4 years)
  Longitudinal medical record data

SECONDARY OUTCOMES:
Change from baseline Obesogenic Behaviors at 2 years | Baseline, 2 year
  Measures include diet (fruit and vegetable consumption, sugar sweetened beverage intake), physical activity, screen time, television in child's bedroom and sleep.
Change from baseline Child Quality of Life at 2 years | Baseline, 2 year
  Measured using scales from the Pediatric Quality of Life Inventory (PedsQL) TM, parent report for child.
Change from baseline Healthcare Satisfaction at 2 years | Baseline, 2 year
  Questions adapted from the Patient Assessment of Chronic Care (PACIC) tool

OTHER OUTCOMES:
Change from baseline Healthcare Utilization at 2 years | Baseline, 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Land, PhD, Principal Investigator — Massachusetts Department of Health; Elsie M Taveras, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Community Health Connections, Inc., Fitchburg, Massachusetts
  - Greater New Bedford Community Health Center, New Bedford, Massachusetts

REFERENCES:
- [Derived] Taveras EM, Perkins M, Anand S, Woo Baidal JA, Nelson CC, Kamdar N, Kwass JA, Gortmaker SL, Barrett JL, Davison KK, Land T. Clinical effectiveness of the massachusetts childhood obesity research demonstration initiative among low-income children. Obesity (Silver Spring). 2017 Jul;25(7):1159-1166. doi: 10.1002/oby.21866. PMID 28653504
- [Derived] Franckle RL, Falbe J, Gortmaker S, Barrett JL, Giles C, Ganter C, Blaine RE, Buszkiewicz J, Taveras EM, Kwass JA, Land T, Davison KK. Student obesity prevalence and behavioral outcomes for the massachusetts childhood obesity research demonstration project. Obesity (Silver Spring). 2017 Jul;25(7):1175-1182. doi: 10.1002/oby.21867. PMID 28653502
- [Derived] Woo Baidal JA, Nelson CC, Perkins M, Colchamiro R, Leung-Strle P, Kwass JA, Gortmaker SL, Davison KK, Taveras EM. Childhood obesity prevention in the women, infants, and children program: Outcomes of the MA-CORD study. Obesity (Silver Spring). 2017 Jul;25(7):1167-1174. doi: 10.1002/oby.21865. PMID 28653498